CLINICAL TRIAL: NCT00888017
Title: Proton Pump Inhibitor Therapy and Bone Density in Premature Infants
Acronym: PPI
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment
Sponsor: University of Utah (Other)
Responsible Party: Gary M Chan, MD, University of Utah
Other Study IDs: 29104
Record Dates: First submitted 2009-04-08; First posted 2009-04-24 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Osteopenia; Prematurity
Keywords: bone density; proton pump inhibitors; premature infants
MeSH Terms: conditions — Bone Diseases, Metabolic; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PPI group: This group of infants have received treatment with a PPI as ordered by their neonatologist during their hospital stay.
- non-PPI group: These infants did not receive PPIs during their hospital stay.

SUMMARY:
Previous research studies have shown that there may be a connection between proton pump inhibitor therapies and hip fracture in adults(1). Proton pump inhibitor(PPI) reflux medications raise the pH of the stomach, which may effect the body's ability to absorb certain calcium compounds.

Neonates are at a crucial age for bone mineralization. Because esophageal reflux is common in neonates, PPI therapy is commonly used, despite little information on effectiveness and side effects. PPIs work by blocking the production of protons in the pumps in the stomach, thus making the stomach less acidic. The calcium ion needs an acidic environment in order to be broken down from its natural compounds into an absorbable form (2). This is troubling because of the problems associated with osteopenia in neonates. Bone mineralization is important for premature infants. Rickets and bone fractures are higher in preterm infants than term infants. For this reason, we are investigating whether there is a connection between PPI therapies (specifically Prevacid) and decreased bone densities in neonates.

The objective is to determine if a connection exists between proton pump inhibitor antacids and decreased rate of bone mineralization in neonates.

DETAILED DESCRIPTION:
After a patient is screened and consent is obtained, participants will all be initially placed into group one. Patients will be later moved to group two if their treatment includes proton pump inhibitors.

Group 1: Patients that meet the selection criteria that are not currently receiving any treatments for reflux or have other excluding conditions.

Group 2: Patients that meet the selection criteria and are receiving proton pump inhibitors as part of their treatment in the NBICU.

Participants in both groups will receive a bone density ultrasound when they begin full feeds, and every two weeks following until discharge. Participants will not be asked to participate in scans post discharge.

Because most babies do not begin GER therapy until some time after they have reached full feedings, they will be placed in group two retrospectively.

During each participating infant's hospital stay, the following procedures will be performed:

Each infant will undergo all of the tests and procedures that would normally be done for his/her care including physical exams, vital signs, and monitoring respiratory status.

Each infant will be weighed and and his/her length and head circumference will also be measured. This is also standard of care.

After the initial scan, each participating infant will receive subsequent bone density ultrasounds once every two weeks until time of discharge. These bone ultrasounds are done by study personnel and will not be charged to the patient or the patient's insurance.

The medications being evaluated in this study are not experimental. Patient care is to the discretion of the treating physician. Standard of care and treatment will not be affected by this study. The only procedures included in this study that are not a standard of care are bone ultrasounds, three weeks apart (number of ultrasounds depends on discharge, death, and other excluding criteria).

ELIGIBILITY:
Inclusion Criteria:

* Infants born between 24 and 34 weeks gestation and 600g to 2000g birth weight Parental consent has been obtained

Exclusion Criteria:

* Infants with bone disorders, liver or kidney problems, infants of diabetics, growth retarded infants, or infants taking diuretics or chronic steroids will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants born between 24 and 34 weeks gestation and 600g to 2000g birth weight.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To determine if a connection exists between proton pump inhibitor antacids and decreased rate of bone mineralization in neonates. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Chan, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Ivanovich P, Fellows H, Rich C. The absorption of calcium carbonate. Ann Intern Med. 1967 May;66(5):917-23. doi: 10.7326/0003-4819-66-5-917. No abstract available. PMID 6025232
- [Result] Yang YX, Lewis JD, Epstein S, Metz DC. Long-term proton pump inhibitor therapy and risk of hip fracture. JAMA. 2006 Dec 27;296(24):2947-53. doi: 10.1001/jama.296.24.2947. PMID 17190895